CLINICAL TRIAL: NCT02920112
Title: Telephone-Based Cognitive Behavioural Therapy for Bariatric Surgery Patients One Year Following Bariatric Surgery: A Pilot Study
Brief Title: Tele-CBT One Year Following Bariatric Surgery: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sanjeev Sockalingam, Deputy Psychiatrist-in-Chief, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0622-BE2; Grant #317877 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2016-09-08; First posted 2016-09-30 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery; Bariatrics; Cognitive Therapy; Binge eating
MeSH Terms: conditions — Obesity; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One year post-op Tele-CBT (Experimental): This group will receive Telephone based Cognitive Behavioral Therapy (Tele-CBT) one year after bariatric surgery.
  Interventions: Behavioral: Telephone based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Telephone based Cognitive Behavioral Therapy — 6 sessions of Telephone based Cognitive Behavioral Therapy over the telephone, lasting approximately 60 minutes each.
  Other Names: Tele-CBT

SUMMARY:
This second phase of a pilot study (non-drug) will examine the effectiveness and feasibility of Telephone based Cognitive Behavioural Therapy (Tele-CBT) as an additional treatment to the usual standard of care in bariatric surgery patients. Participants one year post-surgery will receive six sessions of Tele-CBT and complete measures before, during, immediately after, and one year after participation in the study.

DETAILED DESCRIPTION:
Obesity is an increasingly prevalent chronic condition (Ogden et al., 2006) which is associated with significant health consequences, including type 2 diabetes, obstructive sleep apnea, hypertension, and hyperlipidemia (Bray, 2004). Bariatric surgery is the most effective treatment for patients with extreme obesity (Colquitt et al., 2005). Unfortunately, it has been estimated that 20 to 50% of patients begin to regain their weight within the first 1 ½ to 2 years, and improvements in medical comorbidities dissipate with weight regain (Hsu et al., 1998; Shah et al., 2006). In light of the high relapse rates following bariatric surgery, research on non-surgical factors that influence the outcome of bariatric surgery, such as psychiatric comorbidity, has become increasingly important (Hsu et al., 1998). Up to 55% of bariatric surgery candidates have an Axis I disorder at the time of the initial assessment, with the most common diagnoses being eating disorders (37%), affective disorders (32%), and anxiety disorders (15%) (Muhlhans et al., 2009). Despite accumulating evidence indicating that psychiatric comorbidity is associated with poorer surgical outcomes, psychological interventions are not routinely offered in Bariatric Surgery programs. It has been suggested that cognitive behavioural therapy (CBT) could be helpful in maintaining weight loss (Kalarchian & Marcus, 2003). We have published a paper on the feasibility of the protocol using a small sample and producing promising eating improvements post-intervention (Cassin et al., 2013). A more recent study (Cassin et al., 2016) of the first phase of this study with Tele-CBT delivered 6 months before surgery indicated significant improvements in binge eating, emotional eating, and depressive symptoms, compared to a control group. These results are similar to other studies employing CBT for bariatric surgery patients (e.g. Gade et al., 2014). We have recently published on the outcomes for Tele-CBT delivered 6 months post-surgery (Sockalingam, Cassin, Wnuk, Du, Jackson, Hawa, & Parikh, 2016) that showed significant reductions in scores of binge eating, emotional eating, depression, and anxiety. The same measures used in the first phase of the study (Cassin et al., 2016; Sockalingam et al., 2016) will be used in this second phase, looking at Tele-CBT delivered to patients at one year after surgery. Comparisons between the efficacy of Tele-CBT based on responses to measures will be made for participants receiving the intervention at 6 months before surgery, 6 months after surgery, and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English.
2. Have access to a telephone and a computer with internet connection.
3. Have the capacity to provide informed consent.
4. Patient is at approximately one year post-surgery at the Bariatric Surgery Program at Toronto Western Hospital.

Exclusion Criteria:

1. Active suicidal ideation.
2. Active serious mental illness
3. Active severe depression
4. Active severe anxiety
5. Active symptoms of post-traumatic stress disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Changes in Eating Pathology: Emotional Eating Scale (EES) | Baseline pre-intervention, weekly up to 6 weeks during intervention, immediately post-intervention, and 1 year after intervention,
  25-item self-report measure that assesses tendency to cope with negative affect by eating.
Changes in Eating Pathology: Binge Eating Scale (BES) | Baseline pre-intervention, immediately post-intervention, and 1 year after intervention
Changes in Eating Pathology: Eating Disorder Examination Questionnaire (EDEQ) | Baseline pre-intervention, immediately post-intervention, and 1 year after intervention
  41-item self-report measure that assesses eating disorder psychopathology. Only 3 items regarding binge eating will be used. Will be used to measure changes in eating pathology.
Changes in Eating Pathology: Ontario Bariatric Eating Self-Efficacy Scale (OBESE) - Changes in Eating Pathology | Baseline pre-intervention, immediately post-intervention, and 1 year after intervention
  28-item self-report measure of eating self-efficacy in bariatric patients.

SECONDARY OUTCOMES:
Satisfaction with Therapy: Working Alliance Inventory - Short Form (WAI-SF) | Weekly up to 6 weeks during intervention and immediately post-intervention
  12-item self-report measure that assesses the alliance between patient and therapist.
Changes in Depression Severity | Baseline pre-intervention, weekly up to 6 weeks during intervention, immediately post-intervention, and 1 year after intervention
  Measured with Patient Health Questionnaire (PHQ-9), a 9-item self-report measure of depression severity.
Changes in Anxiety Severity | Baseline pre-intervention, immediately post-intervention, and 1 year after intervention
  Measured with Generalized Anxiety Disorder Questionnaire (GAD-7), a 7-item self-report measure of anxiety severity.
Changes in Health-Related Quality of Life | Baseline pre-intervention, immediately post-intervention, and 1 year after intervention
  Measured with Short-Form Health Survey (SF-36), a 36-item self-report measure of health-related quality of life.
Satisfaction with Therapy: Tele-CBT Client Change Interview | Weekly up to 6 weeks during intervention, immediately post-intervention, 1 year after intervention
  a 9-item self-report measure that qualitatively assesses patient experience with the Tele-CBT treatment
Satisfaction with Therapy: Helpful Aspects of Therapy Form (HAT) | Weekly up to 6 weeks during intervention and immediately post-intervention
  brief, open-ended questionnaire completed by participants after each session. Participants are asked to describe in their own words the most helpful event in the session, and to rate how helpful it was.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Sockalingam, MD, FRCPC, Principal Investigator — University of Toronto, Toronto Western Hospital; Stephanie E Cassin, PhD, CPsych, Principal Investigator — Toronto Metropolitan University; Raed Hawa, MD, FRCPC, Study Director — University of Toronto, Toronto Western Hospital; Susan Wnuk, PhD, CPsych, Study Director — University of Toronto, Toronto Western Hospital; Timothy Jackson, MD, FRCSC, Study Director — University of Toronto, Toronto Western Hospital; Chau Du, MSc, Study Director — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital with the University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly in order to protect patient confidentiality. Aggregate and anonymous data will be shared in peer-reviewed journal articles and scientific presentations.

REFERENCES:
- [Background] Cassin SE, Sockalingam S, Du C, Wnuk S, Hawa R, Parikh SV. A pilot randomized controlled trial of telephone-based cognitive behavioural therapy for preoperative bariatric surgery patients. Behav Res Ther. 2016 May;80:17-22. doi: 10.1016/j.brat.2016.03.001. Epub 2016 Mar 10. PMID 26990279
- [Background] Cassin SE, Sockalingam S, Wnuk S, Strimas R, Royal S, Hawa R, Parikh SV. Cognitive Behavioral Therapy for Bariatric Surgery Patients: Preliminary Evidence for Feasibility, Acceptability, and Effectiveness. Cognitive and Behavioral Practice 20(4): 529-543, 2013.
- [Background] Sockalingam S, Cassin SE, Wnuk S, Du C, Jackson T, Hawa R, Parikh SV. A Pilot Study on Telephone Cognitive Behavioral Therapy for Patients Six-Months Post-Bariatric Surgery. Obes Surg. 2017 Mar;27(3):670-675. doi: 10.1007/s11695-016-2322-x. PMID 27491293
- [Derived] Santiago VA, Cassin SE, Wnuk S, Du C, Hawa R, Parikh SV, Sockalingam S. "If you're offered help, take it": A qualitative study examining bariatric patients' experience of telephone-based cognitive behavioural therapy. Clin Obes. 2021 Apr;11(2):e12431. doi: 10.1111/cob.12431. Epub 2020 Nov 29. PMID 33251753
- [Derived] Sockalingam S, Leung SE, Hawa R, Wnuk S, Parikh SV, Jackson T, Cassin SE. Telephone-based cognitive behavioural therapy for female patients 1-year post-bariatric surgery: A pilot study. Obes Res Clin Pract. 2019 Sep-Oct;13(5):499-504. doi: 10.1016/j.orcp.2019.07.003. Epub 2019 Aug 10. PMID 31409544